CLINICAL TRIAL: NCT06799702
Title: Trauma-informed, Resilience-based Telehealth Intervention for Improving HIV Prevention and HCV Care for Persons Who Inject Drugs in the Deep South
Brief Title: Trauma-informed, Resilience-based Telehealth Intervention for Improving HIV Prevention and HCV Care for Persons Who Inject Drugs in the Deep South (Pilot Testing: Aim3)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mohammad Rifat Haider, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PROJECT000009015; K01DA059329 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HIV Pre-exposure Prophylaxis; HEPATITIS C (HCV); Opioid Use Disorder
Keywords: HIV Pre-Exposure Prophylaxis; Hepatitis C Virus; Medications for Opioid Use Disorder; People who inject drugs (PWID); Deep South; Telehealth Intervention
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention
  Interventions: Behavioral: Telehealth Behavioral Intervention for promoting HIV and HCV care and MOUD among Persons who inject drugs (PWID)
- Waitlist Control (Active Comparator): Control
  Interventions: Behavioral: Telehealth Behavioral Intervention for promoting HIV and HCV care and MOUD among Persons who inject drugs (PWID)

INTERVENTIONS:
Behavioral: Telehealth Behavioral Intervention for promoting HIV and HCV care and MOUD among Persons who inject drugs (PWID) — The telehealth intervention will include components from the LIFT intervention: identifying and expressing emotion related to stressors; identifying different stressors and coping difficulties; and developing adaptive strategies to reduce stress. The intervention will also include developing health goals and a health plan on PrEP, DAA, and MOUD, as well as components from RISE-UP: baseline assessment of individual assets (e.
  g., self-esteem, emotion regulation, positive future orientation), coping with addictive behavior (stress reduction, avoiding unsafe sexual and injection practices, self-care), building relationships (with peers, family, provider), and social support (finding and seeking social support). It will consist of 8 sessions (4 addressing stress and 4 addressing stigma). Each session will last an hour and be conducted weekly for eight consecutive weeks.

SUMMARY:
Evaluate the feasibility, acceptability, and usability of the intervention (primary outcomes) and coping skills and resilience (secondary outcomes) of the telehealth intervention over two months (8 weekly sessions) in a waitlist-controlled, randomized pilot trial using a cross-over design among 40 PWID. The primary outcomes will be feasibility, acceptability, and usability of the intervention. Secondary outcomes will be increased coping skills and resilience, which in turn, will increase status neutral HIV and HCV care and MOUD uptake (longer-term outcomes). Outcomes will be assessed using pre- and post-intervention surveys.

DETAILED DESCRIPTION:
The telehealth intervention will include components from the LIFT intervention: identifying and expressing emotion related to stressors; identifying different stressors and coping difficulties; and developing adaptive strategies to reduce stress. The intervention will also include developing health goals and a health plan on PrEP, DAA, and MOUD, as well as components from RISE-UP: baseline assessment of individual assets (e.g., self-esteem, emotion regulation, positive future orientation), coping with addictive behavior (stress reduction, avoiding unsafe sexual and injection practices, self-care), building relationships (with peers, family, provider), and social support (finding and seeking social support). It will consist of 8 sessions (4 addressing stress and 4 addressing stigma). Each session will last an hour and be conducted weekly for eight consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* People who actively inject drugs verified by visible injection stigmata (needle tracks)
* HIV negative
* Adult (≥18 years)
* lives in rural areas

Exclusion Criteria:

* Living with HIV
* Lives in urban areas
* Not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Months 31-60
  Feasibility of the telehealth intervention will be assessed during baseline, at 2-months, and 4-months among both PWID and interventionists. Feasibility will be assessed by the completion rates of the interventionist training sessions and the participation/drop-out rates of the PWID.
Acceptability of the telehealth intervention | Months 31-60
  Acceptability of the telehealth intervention will be assessed during baseline, at 2-months, and 4-months among both PWID and interventionists. Acceptability will be examined by Likert scale like responses, e.g., "convenient," "a nuisance," "easy to use," and "time-consuming."
Usability of the telehealth intervention | Months 31-60
  Usability of the telehealth intervention will be assessed during baseline, at 2-months, and 4-months among both PWID and interventionists. Usability will be assessed with the USE questionnaire, which captures the perceived usefulness, satisfaction, and ease of use.

SECONDARY OUTCOMES:
Depressive symptoms | Months 31-60
  The Center for Epidemiologic Studies Depression (CES-D) Scale (20 items) will be used to measure depressive symptoms. CES-D Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Resilience | Months 31-60
  The 10-item Connor-Davidson Resilience Scale (CD-RISC) scale will be used to measure resilience. Scores range from 0-40, where higher scores indicate greater resilience.
Intersecting stigma of HIV, HCV, and drug use | Months 31-60
  The 16-item Anticipated HIV Stigma Scale will be used to measure HIV stigma. Scores range from 16-64, where higher scores reflect higher stigma. The 33-item HCV Stigma Scale (HCV-SS) will be used to measure HCV-related stigma. The total score range for this scale is 33 to 132, with higher scores indicating greater perceived stigma. The 8-item Perceived Stigma of Substance Abuse Scale (PSAS) will be used to measure the drug use stigma. Scores range from 8-32, where a higher score reflects higher stigma. Intersectional stigma scores will be calculated using the formula, d = square root of (a-squared + b-squared + c-squared), where d is the intersectional stigma score, and a is the HIV-related stigma score, b is the HCV-related stigma score, and c is the drug use stigma score. The score ranges from 37.5-150.2, and the higher the score, the higher the intersecting stigma.
Sexual behavior | Months 31-60
  Sexual practices like protected sex, risky sex (sex under the influence, sex in return of drugs/money, unprotected anal/vaginal sex, multiple partners, not knowing partnmer's HIV status)
Risky Injection Bheavior | Months 31-60
  Risky injection behavior includes the sharing of syringes, using same syringe multiple times

CONTACTS AND LOCATIONS:
Locations (1):
- MedLink Georgia, Colbert, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Investigators will not share the IPD of the participants of this study due to the risk of privacy breach for the participants.